CLINICAL TRIAL: NCT03941977
Title: Treatment of Bone Marrow Edema Lesions of the Knee With Percutaneous Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 37392614.9.0000.0068
Record Dates: First submitted 2017-02-20; First posted 2019-05-08 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-04

CONDITIONS: Bone Marrow Edema
MeSH Terms: interventions — Magnetic Resonance Imaging; Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery (Experimental): Group evaluated with MRI and submitted to the percutaneous introduction of cannula for bone grafting
  Interventions: Device: Percutaneous introduction of cannula; Diagnostic Test: Magnetic resonance imaging; Biological: Bone Grafting

INTERVENTIONS:
Device: Percutaneous introduction of cannula — An 8 gauge cannula is introduced at the site of the bone marrow lesion. The introduction of the cannula is guided by fluoroscopy.
  Other Names: Arm: Experimental: Surgery
Diagnostic Test: Magnetic resonance imaging — MRI scans will be performed on a 1.5 T (Signa Excite HD, GE Healthcare, Waukesha, WI, USA) and a specific knee coil (HD TRKnee 8 Ch High Resolution Knee Array) will be used.
  Other Names: Arm: Experimental: Surgery
Biological: Bone Grafting — A bone substitute consisting of calcium phosphate will be injected through the cannula, previously inserted, filling the area of the bone marrow lesion. GRAFTYS HBS® (Graftys, Aix en Provence, France) will be used.

SUMMARY:
Objective

1. To evaluate the technique of percutaneous grafting with bone substitute in the knee as to its applicability and technical feasibility.
2. Evaluate the results regarding functional improvement and prevention of the evolution of joint cartilage degeneration.

Material and methods Twenty patients from the Knee Group clinic who meet the criteria will be selected.

Magnetic resonance imaging will be analyzed on the PACS server. Through the resonance will be performed evaluation of the size of the bone edema in volume and its proportion in relation to the size of the affected condyle or tibial plateau and the cartilage of the femoro-tibial joint. The lesions will then be mapped in the coronal and sagittal plane.

Radiographs will be taken in antero-posterior, profile, Rosenberg knee and lower limb views.

Evaluation of the patients will be performed by the visual analog pain scale and by the KOOS, IKDC and SF-36v1 indices.

Description of Surgical Technique After the mapping the patient will be submitted to the procedure. The procedure consists in the application of a bone substitute based on injectable calcium phosphate in the area of bone edema previously mapped with the aid of radioscopy to guide. After confirming the proper positioning of the guidewire, a trephine is introduced through which the product will be injected. GRAFTYS HBS® (Graftys, Aix en Provence, France) will be used.

The procedures will be performed in a surgical center, with conventional antisepsis and asepsis techniques and under spinal anesthesia. The patient will be hospitalized and must be discharged on the first postoperative day. After the procedure the patients will be under partial load as tolerated for two weeks with free range of motion and will start physiotherapy after 2 weeks of the procedure. During hospitalization the patient will receive analgesia with intravenous Dipirone 1g every 6 hours associated with Tramadol 100mg intravenously every 8 hours if severe pain. After discharge the patient will receive analgesia with dipyrone 1g orally every 6 hours associated with Tramadol 100mg orally every 8 hours if severe pain, and Tramadol used by the patient was quantified.

Patients will then be re-evaluated at 1, 3, 12, 24 and 48 weeks with the same previous criteria and at 12 months new MRI with the same previous protocol will be performed.

DETAILED DESCRIPTION:
Initial assessment

All the patients included in the study were submitted to the initial evaluation, in which the following exams and scales were performed:

* Magnetic resonance of the affected knee, according to IOTHCFMUSP standard radiology protocol;
* Panoramic radiography of lower limbs to measure limb alignment;
* X-ray in antero-posterior incidence with load and knee profile;
* Functional ranges of subjective IKDC, KOOS and SF-36v1;
* Analog visual pain scale.

Radiographic evaluation and magnetic resonance imaging

The radiographs were evaluated and classified by a specialist radiologist in musculoskeletal, according to the Kellgren-Lawrence classification. The radiographs were not identified as to the moment of accomplishment, before or after the procedure. However, in many cases it was possible to identify signs of the procedure in the image, making the evaluator blind.

In the MRI images, the location of the bone edema was evaluated in relation to the affected bone (femur or tibia) and affected compartment (medial or lateral). The extent of edema divided into three levels according to the percentage of affected area of the coronal section of the femoral condyle or tibial plateau was also evaluated, with grade 1 being less than 25%, grade 2 between 25% and 50%, and grade 3 greater than 75 %. In the subchondral bone was also recorded the presence of fracture line, cysts and impactions / collapses of the articular surface. In the presence of impaction this was measured in millimeters.

Clinical and functional evaluation

The patients were evaluated by the functional scales: KOOS and subjective IKDC. Quality of life was also assessed by the SF-36v1 questionnaire.

Patient follow-up

Patients were followed in outpatient clinics at 1, 3, 6, 12, 24 and 48 weeks after the surgical procedure. Functional scales were repeated in all consultations. The quality of life scale was repeated at 24 and 48 weeks. Radiographs and MRI were repeated after 48 weeks of surgery.

Description of surgical technique

Magnetic resonance imaging of the patients was mapped in the surgical center to define the area of the lesion, as well as planning of the injection site at the center of the lesion, trajectory and cannula entry point. The cannula trajectory was defined by prioritizing an appropriate angle of attack for the entry point and larger distances of intraosseous trajectory, in order to avoid extravasation of the bone substitute through the cannula inlet.

The procedures were performed under spinal anesthesia, in a surgical center. The patients were placed in dorsal decubitus on a radiolucent table, with a cushion below the ipsilateral hip, for better control of the external rotation of the limb and a cushion also under the ipsilateral knee, aiding in the lateral incidence of fluoroscopy, avoiding the overlap of the knee image contralateral.

The material for the procedure was:

* An 8G metal cannula with distal and lateral exit orifice at the tip
* Metal cannula of the cannula with introductory tip with cut
* Metal cannula embolus with blunt tip
* High Flow Disposable Three-Way Infusion Faucet
* Five 1mL syringes with thread at the tip
* One syringe to prepare the Graftys HBS® bone substitute

According to preoperative planning, with the help of fluoroscopy in front and profile incidences, the cannula entry point was demarcated, with the placement of the cannula on the skin. Incisions of 5 mm in length were performed with a n11 scalpel blade at the point of entry into the skin. The cannulae were introduced, with fluoroscopy control, towards the center of the previously determined lesion. The progression was done manually or with the aid of hammer, when greater resistance was found.

During the introduction of the cannula, oblique incidences of fluoroscopy were performed to avoid perforation of the opposing cortex. The introduction of the cannula was performed very carefully when approaching the opposite cortical, with the possibility of using the blunt tip for cannula, making it difficult to perforation of the cortical.

The bone substitute was then prepared by mixing the solid content with the liquid to liquid / pasty state and transferred to 1 ml syringes. Transfer to smaller diameter syringes is important to achieve an injection flow with lower pressure application. The bone substitutes when subjected to higher pressures pass into a separation phase in which the liquid separates from the solid part, making it impossible to deliver the material in the desired area.

The 1 ml syringes were connected to the cannulae already positioned at the site determined for filling. The bone substitute was injected, interleaving the passage of a metal plunger through the cannula, between each syringe. Through the fluoroscopy it was possible to visualize the distribution of the product in the bone marrow, ensuring that the application was according to the mapping of the lesion and controlling the presence of possible extravasations. The amount of product injected was defined by the control of filling the area of the lesion by fluoroscopy. In cases of intra-articular extravasation, the injection was interrupted. After the injection was completed, it was waited 5 minutes before removal of the cannula, to reduce the reflux of the material through the inlet.

Post-operative care

The patients were hospitalized until the day after the procedure. Full load was allowed as tolerated for two weeks, with free range of motion. During hospitalization, patients received analgesia with intravenous dipyrone 1g every 6 hours, associated with intravenous tramadol 100mg every 8 hours if they presented severe pain greater than 7. After discharge, patients received analgesia with dipyrone 1g orally 6 in 6 hours, associated with tramadol 100mg orally every 8 hours, if severe pain, for a week, and the tramadol used by the patient in this period was quantified.

Surgical incision stitches were removed at the first outpatient appointment 1 week after surgery. The patients did not undergo physiotherapy or any type of rehabilitation after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 85 years
* Gender: both genders
* Knee pain for at least 6 months
* Hypercaption lesion in subchondral region of tibial plateau or femoral condyle in T2-weighted magnetic resonance imaging with fat suppression.

Exclusion Criteria:

* Rheumatologic diseases diagnosed in treatment
* Renal insufficiency requiring hemodialysis
* Not ambulatory
* Knee osteoarthrosis with Kellegren / Lawrence classification greater than 3
* Alignment in varus or valgus greater than 8 degrees in relation to the mechanical axis
* Radiographic changes in the femoro-patellar joint associated with symptoms of anterior knee pain

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | Pre-operative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life
Knee injury and Osteoarthritis Outcome Score | 1 week postoperative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life, comparative with pre-optative evaluation
Knee injury and Osteoarthritis Outcome Score | 3 weeks postoperative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life, comparative with pre-optative evaluation
Knee injury and Osteoarthritis Outcome Score | 6 weeks postoperative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life, comparative with pre-optative evaluation
Knee injury and Osteoarthritis Outcome Score | 12 weeks postoperative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life, comparative with pre-optative evaluation
Knee injury and Osteoarthritis Outcome Score | 24 weeks postoperative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life, comparative with pre-optative evaluation
Knee injury and Osteoarthritis Outcome Score | 48 weeks postoperative
  Evatualion of Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life, comparative with pre-optative evaluation
International Knee Documentation Committee | Pre-operative
  knee-specific patient-reported outcome measure
International Knee Documentation Committee | 1 week postoperative
  knee-specific patient-reported outcome measure, comparative with pre-optative evaluation
International Knee Documentation Committee | 3 weeks postoperative
  knee-specific patient-reported outcome measure, comparative with pre-optative evaluation
International Knee Documentation Committee | 6 weeks postoperative
  knee-specific patient-reported outcome measure comparative with pre-optative evaluation
International Knee Documentation Committee | 12 weeks postoperative
  knee-specific patient-reported outcome measure, comparative with pre-optative evaluation
International Knee Documentation Committee | 24 weeks postoperative
  knee-specific patient-reported outcome measure, comparative with pre-optative evaluation
International Knee Documentation Committee | 48 weeks postoperative
  knee-specific patient-reported outcome measure, comparative with pre-optative evaluation
Short Form 36 Health Survey | Pre-operative
  Patient-reported survey of patient health
Short Form 36 Health Survey | 24 weeks postoperative
  Patient-reported survey of patient health, comparative with pre-optative evaluation
Short Form 36 Health Survey | 48 weeks postoperative
  Patient-reported survey of patient health, comparative with pre-optative evaluation
Visual analog scale for Pain | Pre-operative
  Unidimensional measure of pain intensity
Visual analog scale for Pain | 1 Week postoperative
  Unidimensional measure of pain intensity, comparative with pre-optative evaluation
Visual analog scale for Pain | 3 weeks postoperative
  Unidimensional measure of pain intensity, comparative with pre-optative evaluation
Visual analog scale for Pain | 6 weeks postoperative
  Unidimensional measure of pain intensity, comparative with pre-optative evaluation
Visual analog scale for Pain | 12 weeks postoperative
  Unidimensional measure of pain intensity, comparative with pre-optative evaluation
Visual analog scale for Pain | 24 weeks postoperative
  Unidimensional measure of pain intensity, comparative with pre-optative evaluation
Visual analog scale for Pain | 48 weeks postoperative
  Unidimensional measure of pain intensity, comparative with pre-optative evaluation

SECONDARY OUTCOMES:
Edema Volume evaluation | 1 year postoperative
  MRI evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Marco K Demange, PhD, Principal Investigator — Faculty
Locations (1):
- Hospital das Clinicas - University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No